CLINICAL TRIAL: NCT02174354
Title: Methotrexate Polyglutamates as a Marker of Clinical Response and Toxicity in the Treatment of Psoriasis
Acronym: MTXPG
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 11/H0802/7
Record Dates: First submitted 2014-05-22; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Psoriasis Chronic; Injury of Liver
Keywords: Psoriasis; Methotrexate; Methotrexate Polyglutamates; Injury of Liver
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Longitudinal study design. Serum samples will be retained with consent.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Psoriasis: Patients with psoriasis taking methotrexate

SUMMARY:
Methotrexate (MTX) is widely prescribed to treat inflammatory conditions including psoriasis, where it is the recommended first-line systemic therapy in moderate-to-severe disease. Approximately 40% of patients with psoriasis have a sub-optimal response to MTX and a significant number experience side effects that may include deranged liver enzymes. There is currently no validated test to predict how patients with psoriasis will respond to MTX, in terms of disease outcome and/or toxicity, or to guide dose escalation in this group.

DETAILED DESCRIPTION:
Data for this study is drawn from the BSTOP (Biomarkers of Systemic Treatment Outcomes in Psoriasis) cohort. This is a multi-centre, prospective, cohort study to establish clinically relevant biomarkers and pharmacogenetic markers of systemic treatment outcomes in patients with severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with psoriasis
* Taking oral or subcutaneous methotrexate
* Measurement of methotrexate polyglutamates on at least one occasion during therapy.
* Patients who have given written informed consent

Exclusion Criteria:

* Unable to consent
* Not taking methotrexate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with psoriasis taking methotrexate recruited in outpatient dermatology clinics
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2011-01; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Serial erythrocyte methotrexate polyglutamate measurements using high performance liquid chromotography | From 3 months to 5 years after commencing methotrexate
  To determine if there is a correlation between methotrexate polyglutamate concentrations and clinical response measured by Psoriasis Area Severity Index( PASI) in patients on methotrexate monotherapy with psoriasis. This will consider potential confounding factors, including age, gender and dose of MTX

SECONDARY OUTCOMES:
Alanine transaminase (ALT) and Full blood count (FBC) will be used to measure toxicity to methotrexate | 3 months to 5 years after first MTX dose
  To determine if there is an association between MTXPG levels and evidence of hepatotoxicity in patients with psoriasis taking either (1) methotrexate alone or (2) methotrexate in combination with another systemic drug. Evidence of hepatotoxicity will be determined by the use of current gold standard tests.

OTHER OUTCOMES:
A ROC (Receiver Operating Characteristic) curve will be produced in order to define a therapeutic dose range of MTXPG in psoriasis | 3 months to 5 years after first dose of methotrexate
  If a positive correlation is identified between MTXPG levels and clinical response we aim to define a therapeutic dose range of MTXPG.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine H Smith, MD, Principal Investigator — Kings College London and Guys and St Thomas' NHS Foundation Trust
Locations (1):
- King's College London and Guys' and St Thomas' NHS Foundation Trust, London, London, United Kingdom

REFERENCES:
- [Background] Becker ML, Gaedigk R, van Haandel L, Thomas B, Lasky A, Hoeltzel M, Dai H, Stobaugh J, Leeder JS. The effect of genotype on methotrexate polyglutamate variability in juvenile idiopathic arthritis and association with drug response. Arthritis Rheum. 2011 Jan;63(1):276-85. doi: 10.1002/art.30080. PMID 20954192
- [Background] Woolf RT, West SL, Arenas-Hernandez M, Hare N, Peters van Ton AM, Lewis CM, Marinaki AM, Barker JN, Smith CH. Methotrexate polyglutamates as a marker of patient compliance and clinical response in psoriasis: a single-centre prospective study. Br J Dermatol. 2012 Jul;167(1):165-73. doi: 10.1111/j.1365-2133.2012.10881.x. PMID 22309614
- [Background] Stamp LK, O'Donnell JL, Chapman PT, Zhang M, Frampton C, James J, Barclay ML. Determinants of red blood cell methotrexate polyglutamate concentrations in rheumatoid arthritis patients receiving long-term methotrexate treatment. Arthritis Rheum. 2009 Aug;60(8):2248-56. doi: 10.1002/art.24653. PMID 19644853